CLINICAL TRIAL: NCT01850732
Title: Screening of Abdominal Aortic Aneurysms Among Male Patients With TIA Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Vänni, General surgeon, North Karelia Central Hospital
Purpose: Screening
Other Study IDs: AAA-03
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound of aorta (Other)
  Interventions: Other: Ultrasound of aorta

INTERVENTIONS:
Other: Ultrasound of aorta

SUMMARY:
The purpose of this study is to investigate the prevalence of abdominal aortic aneurysms (AAA) among male patients with transient ischemic attack (TIA) symptoms. Ethiology of AAA is known to be common with atherosclerotic arterial diseases (coronary artery disease, peripheral artery disease and carotid artery disease), so the hypothesis is that AAA should be more common among these TIA patients, thus making screening of these patients (for AAA) more cost-efficient.

Study will be carried out as a prospective screening study. Data will be collected in North Karelia Central Hospital within one year. All male patients with TIA symptoms will be recruited for the study and screened for AAA with ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* male patient who has had symptoms of transient ischemic attack (TIA)

Exclusion Criteria:

* Patient's denial to participate
* Female gender
* Already diagnosed or treated abdominal aortic aneurysm

Sex: Male
Age Groups: Child, Adult, Older Adult
Dates: Start 2013-05; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum diameter (mm) of abdominal aorta (outer-to-outer wall) in ultrasound | upon screening (collection of data will take one year)

CONTACTS AND LOCATIONS:
Locations (1):
- North Carelia Central Hospital, Joensuu, Pohjois-Karjala, Finland